CLINICAL TRIAL: NCT05881928
Title: Effect of Adding Lamotrigine to Sodium Valproate in Childhood Epilepsy: Clinicolabratory Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdellatief, Principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: lamotrigine , sodium valproate
Record Dates: First submitted 2023-03-21; First posted 2023-05-31 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy; Lamotrigine; Sodium Valproate Adverse Reaction
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid; Lamotrigine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 50 epileptic patients receive SV for 6 months , for whom add lamotrigine for 6 month (Other): 50 epileptic patients receive SV for 6 months at dose 30 mg.kg.day, for whom add lamotrigine for 6 month at dose 0.5 mg.kg.day then add 0.5 mg.kg.day every 2 weeks
  Interventions: Drug: Sodium Valproate 500 Mg Prolonged-Release Oral Tablet; Drug: Lamotrigine; Device: E.E.G

INTERVENTIONS:
Drug: Sodium Valproate 500 Mg Prolonged-Release Oral Tablet — sodium valproate tablet30 mg / kg / day , maximum 1500mg / day . LTG :
Drug: Lamotrigine — lamotrigine tablet 0.5 mg/kg for 2 weeks in two divided doses , increased in 0.5mg/kg/day increments every 2weeks .
Device: E.E.G — device recording of brain activity. During this painless test, small sensors are attached to the scalp to pick up the electrical signals produced by the brain. These signals are recorded by a machine and are looked at by a doctoris

SUMMARY:
Epilepsy is one of the most common serious chronic brain disorders of childhood. The causes of epilepsy include :acquired brain damage, altered metabolic states, inborn brain malformations, and genetic causes. At present, antiepileptic drugs (AEDs) are the first line therapy for resistant epilepsy (RE) , and the second line is surgery , and vagus nerve stimulation . Sodium valproate (SV) is a first line anti epileptic drug that can be applied to various seizure types in children . SV has anticonvulsant activity through regulation of neuronal pathways . It has a molecular structure similar to neurotransmitter γ aminobutyric acid (GABA) resulting in GABA synergism , A serious adverse effect of the valproic acid (VPA) : is its effect on liver function with resultant drug-induced hepatotoxicity, hyperammonemia . Lamotrigine (LTG) is a second generation AED

. LTG belongs to the sodium channel blocking class of antiseizure medications (ASMs). Lamortigine side effects include severe rash, fever, lymphadenopathy, hepatic dysfunction, blood disorder,and disseminated intravascular coagulation and Stevens-Johnson syndrome (SJS) . the aim : Evaluation of the efficacy and safety of adding lamotrigine to sodium valproate in epileptic children not responding to SV alone for 6 months. Moreover, the investigators will evaluate the effects of this addition ,appearance of side effects,laboratory evaluation and EEG changes 50 epileptic patients receive SV for 6 months without complete remission for participants, the investigators will add lamotrigine for 6 months.

DETAILED DESCRIPTION:
Epilepsy is one of the most common serious chronic brain disorders of childhood. It is characterized by recurrent seizures that can cause motor, sensory, cognitive, psychic, or autonomic disturbances. It has a negative impact on 0.6% of the population in developed countries and 1.6% in developing countries . The causes of epilepsy include :acquired brain damage, altered metabolic states, inborn brain malformations, and genetic causes .. At present, antiepileptic drugs (AEDs) are the first line therapy for resistant epilepsy (RE) , and the second line is surgery , and vagus nerve stimulation . Although the treatment for RE has been continuously updated, the exploration of high efficacy AED combinations is still ongoing . Sodium valproate (SV) is a first line anti epileptic drug that can be applied to various seizure types in children . SV has anticonvulsant activity through regulation of neuronal pathways . It has a molecular structure similar to neurotransmitter γ aminobutyric acid (GABA) resulting in GABA synergism , A serious adverse effect of the valproic acid (VPA) : is its effect on liver function with resultant drug-induced hepatotoxicity, hyperammonemia . Lamotrigine (LTG) is a second generation AED , and also has the function of resisting depression and stabilizing mood . It is applicable for children and adolescents with various seizure types and syndromes due to its good anticonvulsant, tolerance, broad spectrum activity, and safety . LTG belongs to the sodium channel blocking class of antiseizure medications (ASMs). Lamortigine side effects include severe rash, fever, lymphadenopathy, hepatic dysfunction, blood disorder,and disseminated intravascular coagulation and Stevens-Johnson syndrome (SJS) has also been mentioned as a rare hypersensitivity reaction . The aim : Evaluation of the efficacy and safety of adding lamotrigine to sodium valproate in epileptic children not responding to SV alone for 6 months. Moreover, the investigators will evaluate the effects of this addition ,appearance of side effects,laboratory evaluation and EEG changes 50 epileptic patients receive SV for 6 months without complete remission for participants, Investigators will add lamotrigine for 6 months. Setting: single -center study with outpatient from University Children's Hospital , Faculty of Medicine , Assuit University Design of this study :- Cross -sectional interventional. Selected patient for this study will receive additional treatment of LTG with SV for 6 month .

Doses of the drugs: Sodium valproate : 30 mg / kg / day , maximum dose 1500mg / day . LTG will be initiated at a daily dose of 0.5 mg/kg for 2 weeks in two divided doses, followed by 1.0 mg/kg/day for an additional 2 weeks,followed by 1.5mg/kg/day for additional 2weeks Thereafter, doses will be increased in 0.5mg/kg/day increments every 2weeks until intolerable adverse effects occurred, or a maximum dose of 3mg/kg/day will be reached .

The outcome measures :

The outcome measures will be . 1.Clinical measures: -patient will be clinically examined For side effects(body weight ,muscle weakness ,ataxia , hair loss). - The seizure frequency before and after adding lamotrigine. the investigators will exclude patient with allergy to LTG after the first 2 weeks of treatment.

2- Laboratory measures :- -Serum concentration of lamotrigine at the end of study . - The incidence of adverse reactions will be assessed by lab tests as 1. liver function tests. 2.serum ammonia 3. coagulation function 4. complete blood count. 3-Neurophysological evaluation:-EEG will be done at the beginning and end of the study.

Inclusion criteria : 1. Male or female, ages 2 - 12years.

2 . 50 epileptic children on sodium valproate for 6 months without complete remission.

Exclusion Criteria:

Subjects will be excluded if any of the following criteria are met:-

1. Suspected other neurological disorders .
2. Allergic to LTG.
3. Liver dysfunction.
4. kidney dysfunction .
5. Not cooperating with this study

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 2 - 12years.
* 50 epileptic children on sodium valproate for 6 months without complete remission.

Exclusion Criteria:

* other neurological disorders .
* Allergic to LTG.
* Liver dysfunction.
* kidney dysfunction .
* Not cooperating with this study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-07-29 (Estimated); Primary Completion 2024-07-30 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Weight | 6 months
  Weight in kilogramme will be measured in 50 participants

SECONDARY OUTCOMES:
liver function tests | 6months
  blood tests that measure different enzymes, proteins, and other substances made by the liver.The liver function tests typically include alanine transaminase (ALT) and aspartate transaminase (AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), serum bilirubin, prothrombin time (PT), the international normalized ratio (INR), total protein and albuminALT. 7 to 55 units per liter (U/L) AST. 8 to 48 U/L. ALP. 40 to 129 U/L. Albumin. 3.5 to 5.0 grams per deciliter (g/dL) Total protein. 6.3 to 7.9 g/dL. Bilirubin. 0.1 to 1.2 milligrams per deciliter (mg/dL) GGT. 8 to 61 U/L. LD. 122 to 222 U/L.
serum ammonia. | 6months
  An ammonia test measures the amount of ammonia in the blood , Ammonia level normal range is usually :
  170-340 mcg/dL in new-borns, 70-135 mcg/dL in children , Ammonia Colorimetric Assay Kit will be used for assessment of serum ammonia levels
complete blood count | 6 months
  complete blood count, or CBC, is a blood test that measures many different parts and features of blood, including red blood cells, white blood cells, and platelets
E.E.G | 6months
  E.E.G power in alpha band ,device recording of brain activity. During this painless test, small sensors are attached to the scalp to pick up the electrical signals produced by the brain. These signals are recorded by a machine and are looked at by a doctorisThe most commonly studied waveforms include delta (0.5 to 4Hz); theta (4 to 7Hz); alpha (8 to 12Hz); sigma (12 to 16Hz) and beta (13 to 30Hz). In addition, there are other waveforms such as infra slow oscillations (ISO) (less than 0.5Hz) and high-frequency oscillations (HFOs) (greater than 30Hz) which are outside the conventional bandwidth of clinical EEG but have recently found clinical importance with the adven
Serum concentration of LTG | 6 months
  The serum concentration should be interpreted in the context of the patient's clinical response and may provide useful information in patients showing poor response, noncompliance, or adverse effects, particularly when lamotrigine is coadministered with other epileptic drugs.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altunbasak S, Baytok V, Tasouji M, Herguner O, Burgut R, Kayrin L. Asymptomatic hyperammonemia in children treated with valproic acid. J Child Neurol. 1997 Oct;12(7):461-3. doi: 10.1177/088307389701200709. No abstract available. PMID 9373804
- [Background] Armeno M, Verini A, Del Pino M, Araujo MB, Mestre G, Reyes G, Caraballo RH. A Prospective Study on Changes in Nutritional Status and Growth Following Two Years of Ketogenic Diet (KD) Therapy in Children with Refractory Epilepsy. Nutrients. 2019 Jul 14;11(7):1596. doi: 10.3390/nu11071596. PMID 31337135
- [Background] Balagura G, Iapadre G, Verrotti A, Striano P. Moving beyond sodium valproate: choosing the right anti-epileptic drug in children. Expert Opin Pharmacother. 2019 Aug;20(12):1449-1456. doi: 10.1080/14656566.2019.1617850. Epub 2019 May 17. PMID 31099271
- [Background] Cavus I, Romanyshyn JC, Kennard JT, Farooque P, Williamson A, Eid T, Spencer SS, Duckrow R, Dziura J, Spencer DD. Elevated basal glutamate and unchanged glutamine and GABA in refractory epilepsy: Microdialysis study of 79 patients at the yale epilepsy surgery program. Ann Neurol. 2016 Jul;80(1):35-45. doi: 10.1002/ana.24673. Epub 2016 Jun 13. PMID 27129611
- [Background] Fassi G, Igoa A, Liste OA. [Valproate-induced hyperammonemic encephalopathy. Review of cases in the psychiatric setting]. Vertex. 2008 Nov-Dec;19(82):371-7. Spanish. PMID 19424520
- [Background] Deng J, Fu ZR, Wang L, Liu J, Chen CH, Fang F, Wang XL. Acute liver failure associated with lamotrigine in children with epilepsy: A report of two cases and thoughts on pharmacogenomics. Epilepsy Behav Rep. 2022 Oct 19;20:100568. doi: 10.1016/j.ebr.2022.100568. eCollection 2022. PMID 36345310
- [Background] Fu J, Peng L, Wang W, He H, Zeng S, Chen TC, Chen Y. Sodium Valproate Reduces Neuronal Apoptosis in Acute Pentylenetetrzole-Induced Seizures via Inhibiting ER Stress. Neurochem Res. 2019 Nov;44(11):2517-2526. doi: 10.1007/s11064-019-02870-w. Epub 2019 Sep 11. PMID 31512113
- [Background] Lheureux PE, Hantson P. Carnitine in the treatment of valproic acid-induced toxicity. Clin Toxicol (Phila). 2009 Feb;47(2):101-11. doi: 10.1080/15563650902752376. PMID 19280426
- [Background] Zhang D, Qiu L, Zhang Y, Sang Y, Zheng N, Liu X. Efficacy and safety of sodium valproate plus lamotrigine in children with refractory epilepsy. Exp Ther Med. 2020 Sep;20(3):2698-2704. doi: 10.3892/etm.2020.8984. Epub 2020 Jul 10. PMID 32765764
- [Background] Moosa ANV. Antiepileptic Drug Treatment of Epilepsy in Children. Continuum (Minneap Minn). 2019 Apr;25(2):381-407. doi: 10.1212/CON.0000000000000712. PMID 30921015